CLINICAL TRIAL: NCT04900428
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and Pharmacokinetics of a Single Intranasal Dose of STI-2099 (COVI-DROPS™) in Outpatient Adults With COVID-19
Brief Title: Study to Evaluate a Single Intranasal Dose of STI-2099 (COVI-DROPS™) in Outpatient Adults With COVID-19 (UK)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated at interim analysis due to drops not working on new variants
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRP-COV-201UK
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Covid19
Keywords: covid-19
MeSH Terms: conditions — COVID-19 | interventions — STI-2020

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVI-DROPS (Experimental): 10 mg or 20 mg of COVI-DROPS administered intranasally
  Interventions: Biological: COVI-DROPS
- Placebo (Placebo Comparator): 1 mL administered intranasally
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: COVI-DROPS — COVI-DROPS is a fully human monoclonal antibody which is a neutralizing antibody to SARS-CoV-2
  Other Names: STI-2099
  Arms: COVI-DROPS
Drug: Placebo — Diluent solution
  Arms: Placebo

SUMMARY:
This is a double-blind study designed to investigate the efficacy, safety and PK of a single dose of COVI-DROPS or matched placebo in outpatient adults who have tested positive for COVID-19 and are either asymptomatic or have mild symptoms.

DETAILED DESCRIPTION:
Subjects will be randomized 2:2:1 to receive a single dose of COVI-DROPS 10 mg, COVI-DROPS 20 mg or matched placebo in a double-blind manner. Investigational product (COVI-DROPS or matched placebo) will be administered once as two separate 0.5 mL instillations (0.5 mL up each nostril). Subjects will be followed to Day 60.

ELIGIBILITY:
Inclusion Criteria:

* Positive for COVID-19 with any locally approved RT-PCR within 7 days of planned treatment.
* Either have no COVID-19 symptoms (asymptomatic) or mild illness/symptoms
* Must be willing and able to comply with all planned study procedures and be available for all in-person and telephonic study visits and follow-up as required per protocol
* Subject must have provided written informed consent
* Willing to follow contraception guidelines

Exclusion Criteria:

* Moderate or severe illness/symptoms or rapidly progressive symptoms which are likely to progress such that a hospitalization is imminent (within 24-48 hours)
* Any medical condition that, in the Investigator's opinion, could adversely impact subject safety or key objectives of the study, including any intranasal pathology, or clinically significant laboratory abnormalities, or active clinical disease process
* Documented acute infection other thand COVID-19
* Pregnant or lactating women who are breast feeding or planning to during the study
* Has participated, or is participating, in a clinical research study evaluating COVID-19 convalescent plasma, mAbs against SARS-CoV-2, or intravenous immunoglobulin (IVIG) within 3 months or less than 5 half-lives of the investigational product (whichever is longer) prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Viral load change from baseline to D8 | Baseline to Day 8
  Viral load change from baseline to D8, based on reverse-transcriptase polymerase chain reaction (RT-PCR) determined COVID-19 viral titres (Log-10 copies/mL) from nasopharyngeal swabs

SECONDARY OUTCOMES:
The number of COVID-19-related urgent medically attended visits, emergency department assessments or hospitalizations through D29 | Baseline through Day 29
  The number of COVID-19-related urgent medically attended visits, emergency department assessments or hospitalizations through D29
Proportion of subjects alive and free of hospitalization ˃ 24h duration for acute COVID-19 illness management through D29 | Baseline through Day 29
  Proportion of subjects alive and free of hospitalization ˃ 24h duration for acute COVID-19 illness management through D29
Change in WHO Clinical Progression Scale score | Baseline to Day 8 and Day 29
  Change in WHO Clinical Progression Scale score at D8 and D29 (score of 0-10, with lower score meaning better outcome)
Worst WHO Clinical Progression Scale score up to D8 and from D9 to D29 | Baseline through Day 29
  Worst WHO Clinical Progression Scale score up to D8 and from D9 to D29 (score of 0-10, with lower score meaning better outcome)
Viral load change from baseline to D29 based on RT-PCR determined COVID-19 viral titers (Log-10 copies/mL) from nasopharyngeal swabs | Baseline to Day 29
  Viral load change from baseline to D29 based on RT-PCR determined COVID-19 viral titers (Log-10 copies/mL) from nasopharyngeal swabs
Change in patient-reported COVID-19 symptoms | Baseline to Day 8 and Day 29
  Change in patient-reported COVID-19 symptoms as assessed using the Patient Reported Outcome Instrument for Capture of COVID-19-Related Symptoms (score of 0-50, with lower score meaning better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (1):
- University Hospitals of Coventry and Warwickshire Hospital Trust, Coventry, United Kingdom

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343